CLINICAL TRIAL: NCT02602938
Title: Aspirin on CTCs of Advanced Breast and Colorectal Cancer
Acronym: ACABC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Chao Ni, Dr.Ni, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015KY163
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Epithelial-Mesenchymal Transition; Circulating Tumor Cells
Keywords: aspirin; circulating tumor cells; metastatic breast cancer; metastatic colorectal cancer
MeSH Terms: conditions — Neoplastic Cells, Circulating; Breast Neoplasms; Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- aspirin (Experimental): * The included patients will be administered with aspirin (100mg) orally once a day in 28-day cycles.
  * The CTC was evaluated at baseline, and every 28 days for 2 months.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Take aspirin (100mg) orally once a day for 2 months
  Other Names: acetylsalicylic acid

SUMMARY:
The purpose of this study is to determine whether Aspirin could affect the number and subtype of circulating tumor cells of metastatic breast cancer and colorectal cancer.

DETAILED DESCRIPTION:
BACKGROUND:

* Invasion and metastasis are the main reason of death in metastatic cancer, and abundant evidence find circulating tumor cells(CTCs) take the core position in breast and colorectal cancer metastasis.
* Platelets play multiple role to facilitate the epithelial to mesenchymal transition of tumor cells and protect CTCs to survival in the circulation, which enrolled in the whole process of metastasis.
* Several clinical trials and observational study have validate the primary and secondary prevention effect of aspirin to both breast and colorectal cancer.

OBJECTIVES:

* Determine the effect of aspirin on CTC number of metastatic breast and colorectal cancer;
* Determine the effect of aspirin on CTC subtype (epithelial/mesenchymal/mixed type) of metastatic breast and colorectal cancer.

ELIGIBILITY:

* Adults age from 18-75 years old.
* Patients were diagnosed for metastatic breast or colorectal cancer by pathology.
* Patients who were not currently receiving intravenous chemotherapy , oral administrated with capecitabine was permitted. Concurrent endocrine therapy ( for at least 2 months before enrollment), bisphosphonate therapy, and/or monoclonal targeted therapy were permitted.
* No disease of hemorrhagic tendency or history of non-steroid drug allergy.
* CTCs≥5 / 7.5ml blood

STUDY DESIGN:

* Aspirin will be administered orally once a day in 28-day cycles.
* The CTC was evaluated every 28 days for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults age from 18-75 years old.
* Patients were diagnosed for metastatic breast or colorectal cancer by pathology.
* Patients who were not currently receiving intravenous chemotherapy , oral administrated with capecitabine was permitted.
* Concurrent endocrine therapy ( for at least 2 months before enrollment), bisphosphonate therapy, and/or monoclonal targeted therapy were permitted.
* PS score ≤ 3
* Anticipated survival time ≥ 3 months
* CTCs≥5 / 7.5ml blood

Exclusion Criteria:

* Allergic to aspirin or other types of non-steroid
* History of hemorrhage of digestive tract or other hemorrhagic disease
* Plan to receive surgery within the time frame of the trial
* Medication history of aspirin or other types of anti-platelets drug within one months before the trial
* Women in pregnant or lactation period
* Any psychological or objective problem may influence the compliance of the patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Intervention completed | 2 months
  2-months follow-up completed and the CTCs' assessment was evaluated three times by Canpatrol technology, the tumor burden was evaluated by MRI or CT.

SECONDARY OUTCOMES:
Disease progression | 2 months
  The tumor burden would be examined by MRI or CT once a month, if we find the cancer progressed and chemotherapy is needed, the patient will be withdraw.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang provincial people's hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Ksiazkiewicz M, Markiewicz A, Zaczek AJ. Epithelial-mesenchymal transition: a hallmark in metastasis formation linking circulating tumor cells and cancer stem cells. Pathobiology. 2012;79(4):195-208. doi: 10.1159/000337106. Epub 2012 Apr 4. PMID 22488297
- [Background] Rothwell PM, Wilson M, Price JF, Belch JF, Meade TW, Mehta Z. Effect of daily aspirin on risk of cancer metastasis: a study of incident cancers during randomised controlled trials. Lancet. 2012 Apr 28;379(9826):1591-601. doi: 10.1016/S0140-6736(12)60209-8. Epub 2012 Mar 21. PMID 22440947
- [Background] Maity G, De A, Das A, Banerjee S, Sarkar S, Banerjee SK. Aspirin blocks growth of breast tumor cells and tumor-initiating cells and induces reprogramming factors of mesenchymal to epithelial transition. Lab Invest. 2015 Jul;95(7):702-17. doi: 10.1038/labinvest.2015.49. Epub 2015 Apr 13. PMID 25867761
- [Derived] Yang L, Lv Z, Xia W, Zhang W, Xin Y, Yuan H, Chen Y, Hu X, Lv Y, Xu Q, Weng X, Ni C. The effect of aspirin on circulating tumor cells in metastatic colorectal and breast cancer patients: a phase II trial study. Clin Transl Oncol. 2018 Jul;20(7):912-921. doi: 10.1007/s12094-017-1806-z. Epub 2017 Dec 14. PMID 29243075